CLINICAL TRIAL: NCT06321289
Title: Allogeneic TRAC Locus-inserted CD19-targeting Synthetic T-cell Receptor Antigen Receptor (STAR) T Cells for Relapsed/Refractory B-cell Non-Hodgkin's Lymphoma
Brief Title: Allogeneic TRAC Locus-inserted CD19-targeting STAR T Cell Therapy in r/r B-NHL
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Han weidong, Director of Biotherapeutic Department, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CHN-PLAGH-BT-084
Record Dates: First submitted 2024-03-13; First posted 2024-03-20 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Non-hodgkin Lymphoma,B Cell
MeSH Terms: interventions — fludarabine; fludarabine phosphate; Injections; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Allogeneic TRAC locus-inserted CD19-targeting STAR T cells (Experimental): A conditioning chemotherapy regimen of fludarabine and cyclophosphamide (FC regimen) will be administered followed by investigational treatment, allogeneic targeting CD19 synthetic T-cell receptor antigen receptor T cells.
  Interventions: Biological: Allogeneic CD19-STAR T cell; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Biological: Allogeneic CD19-STAR T cell — Phase 1 dose escalation (3+3): dose 1 (2×10^6 cells/kg), dose 2 (6×10^6 cells/kg), dose 3 (1.8×10^7 cells/kg); Phase 2: dose of RP2D. No more than 5 × 10^4 per kilogram of allogenic residual TCR-positive T cells harbouring in grafts can only be released for recipient infusion.
  Other Names: Allogeneic CD19-targeting synthetic T-cell receptor antigen receptor T cells
Drug: Fludarabine — Intravenous fludarabine 30-50 mg/m^2/day on days -5, -4, and -3.
  Other Names: Fludarabine Phosphate for Injection
Drug: Cyclophosphamide — Intravenous cyclophosphamide 500-1000 mg/m^2/day on days -5, -4, and -3.
  Other Names: Cyclophosphamide for Injection

SUMMARY:
The team has developed the synthetic T cell receptor (TCR) and antigen receptor (STAR) T cells which were demonstrated safety in relapsed or refractory (r/r) B-cell non-Hodgkin' s lymphoma (B-NHL) (NCT05631912). Based on this research, allogeneic STAR-T cell products utilized the CRISPR-Cas9 gene editing tool to knock out endogenous receptor α constant (TRAC), human leukocyte antigen (HLA)-A/B, CIITA, and programmed death 1 (PD-1) genes simultaneously in T cells from healthy donors, and integrated the STAR molecule into the TRAC locus using adenovirus associated virus. This strategy can reduce graft-versus-host-disease (GvHD) toxicity and host-versus-graft response, decrease the sensitivity of STAR T cells to immunosuppressive signals, and improve their anti-tumor activity. In this single center, prospective, open-label, single-arm, phase 1/2 study, the safety and efficacy of allogeneic CD19-targeting STAR T cell therapy will be evaluated in patients with r/r B-NHL.

DETAILED DESCRIPTION:
Phase 1 (dose escalation)

In phase 1, 6 to 18 subjects will be enrolled. Subjects will receive 3 doses of allogeneic CD19-STAR T cell therapy (2 × 10^6 cells/kg, 6 × 10^6 cells/kg, 1.8 × 10^7 cells/kg) from low dose to high dose according to the "3 + 3" principle:

1. Three patients were enrolled in the lowest dose group.
2. Subsequent patients were enrolled according to the following rules:

   1. If the incidence of dose limiting toxicity (DLT) was 0/3, 3 patients were enrolled in the next high-dose group.
   2. If the incidence of DLT was 1/3, 3 patients were enrolled at the same dose; If the incidence of DLT was 1/3 + 0/3, 3 patients were enrolled in the next high-dose group. If the incidence of DLT was 1/3 + 1/3, this dose was defined as maximum tolerated dose (MTD); If the incidence of DLT was 1/3 + 2/3 or 1/3 + 3/3, the previous dose was MTD.
   3. If the incidence of DLT was 2/3 or 3/3, the previous dose was MTD.

To ensure the safety of the subjects, the first subject in each dose group was observed for at least 28 days after the cell infusion. If no DLT occurred, the remaining two subjects could be enrolled and treated at the same dose level. The safety data of all subjects in each dose group until day 28 should be reviewed and tolerated before proceeding to the next dose group trial. No dose escalation was allowed for the same subject during the trial. If a subject drop out during the observation period due to non-DLT reasons, new subjects should be enrolled to make up for the number of subjects who drop out.

Phase 2 (expansion cohort)

In phase 2, 10 to 12 subjects will be enrolled and receive allogeneic CD19-STAR T cell infusion at dose of recommended phase 2 dose (RP2D), which will be determined based on the MTD, occurrence of DLT, the obtained efficacy results, pharmacokinetics / pharmacodynamics and other data according to the phase 1.

Objectives

The primary objectives of the phase 1 are to evaluate the tolerability, safety, and determine RP2D. The primary purpose of the phase 2 study is to evaluate the efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 (inclusive).
2. Patients with histologically confirmed CD19-positive B-cell NHL, including the following types defined by the World Health Organization (WHO) 2016:

   * Diffuse large B-cell lymphoma not otherwise specified (DLBCL-NOS), including activated B-cell type (ABC) / germinal center B-cell Type (GCB);
   * Primary mediastinal (thymic) large B-cell lymphoma (PMBCL);
   * Transformed follicular lymphoma (TFL);
   * High-grade B-cell lymphoma with MYC and BCL2 and/or BCL6 rearrangements (HGBCL);
   * Follicular lymphoma (FL);
   * Mantle cell lymphoma (MCL) [pathologically confirmed, with documentation of monoclonal B cells that have a chromosome translocation t(11;14)(q13;q32) and/or overexpress cyclin D1];
   * Marginal zone lymphoma (MZL), including nodal or splenic marginal zone B-cell lymphoma and mucosa-associated lymphoid tissue (MALT) lymphoma.
3. Relapse after treatment with ≥2 lines systemic therapy for all the above disease types, or refractory disease for aggressive types (DLBCL-NOS, PMBCL, TFL and HGBCL). Relapse disease is defined as disease progression after last regimen. Refractory disease is defined as no CR to first-line therapy:

   * Evaluation of PD (never reached response or SD) after standard first-line treatment, or
   * SD as best response after at least 4 cycles of first-line therapy (eg, 4 cycles of R-CHOP), or
   * PR as best response after at least 6 cycles and biopsy-proven residual disease or disease progression ≤ 6 months of therapy, or
   * Refractory post-autologous stem cell transplant (ASCT): i. Disease progression or relapsed less than or equal to 12 months of ASCT (must have biopsy proven recurrence in relapsed individuals); ii. If salvage therapy is given post-ASCT, the individual must have had no response to or relapsed after the last line of therapy.
4. Individuals must have received adequate prior therapy:

   For MCL, prior therapy must have included:
   * Anthracycline or bendamustine-containing chemotherapy and
   * Anti-CD20 monoclonal antibody (unless investigator determines that tumor is CD20-negative) and
   * Bruton tyrosine kinase inhibitor (BTKi)

   For other types, prior therapy must have included:
   * Anti-CD20 monoclonal antibody (unless investigator determines that tumor is CD20-negative) and
   * Anthracycline containing chemotherapy regimen.

   For individual with TFL must have relapse or refractory disease after transformation to DLBCL.
5. The estimated survival time is over 3 months.
6. The Eastern Cooperative Oncology Group (ECOG) score is 0-2.
7. According to Lugano response criteria 2014, there should be at least one evaluable tumor focus. Evaluable tumor focus was defined as that with the longest diameter of intranodal focus > 1.5cm, the longest diameter of extranodal focus > 1.0cm assessed by computed tomography (CT) or magnetic resonance imaging (MRI).
8. Subjects must be willing to undergo either excised or large-needle lymph node or tissue biopsy, or provide formalin-fixed paraffin-embedded (FFPE) tumor tissue block or freshly cut unstained slides.
9. Functions of important organs meet the following requirements:

   * Echocardiography showed left ventricular ejection fraction ≥50%;
   * Serum creatinine ≤1.5 × upper limit of normal range (ULN) or endogenous creatinine clearance ≥45mL/min (cockcroft-gault formula);
   * Total bilirubin ≤1.5× ULN;
   * Pulmonary function: ≤CTCAE grade 1 dyspnea and oxygen saturation of blood (SaO2) ≥91% in indoor air environment.
10. Blood routine: hemoglobin (Hgb) ≥ 80g/L, neutrophil count (ANC) ≥ 1 × 10 ^ 9/L, platelet count (PLT) ≥ 75 × 10 ^ 9/L. Excluding when there is bone marrow infiltration. It is not allowed to obtain normal values through growth factor intervention.
11. Pregnancy tests for women of childbearing age shall be negative; Both men and women agreed to use effective contraception during treatment and during the subsequent 1 year.
12. Toxicity from previous antitumor therapy ≤ grade 1 (according to CTCAE version 5.0) or to an acceptable level of inclusion/exclusion criteria (other toxicities such as alopecia and vitiligo considered by the investigator to pose no safety risk to the subject).
13. No obvious hereditary diseases.
14. Able to understand the requirements and matters of the trial, and willing to participate in clinical research as required.
15. Informed consent must be signed.

Exclusion Criteria:

1. During the screening period, there was central nervous system (CNS) invasion or a history of clinically significant CNS diseases, such as epilepsy and cerebrovascular diseases.
2. Women who are pregnant or breastfeeding, or who do not agree to use effective contraception during treatment and during the subsequent 1 year.
3. History of allogeneic hematopoietic stem cell transplantation, or organ transplantation.
4. History of other malignancies that have not been in remission.
5. Patients with primary immunodeficiency or autoimmune diseases requiring immunosuppressive therapy.
6. Received radiotherapy within 3 months before enrollment.
7. Received immunotherapy drugs within 4 weeks before enrollment, such as anti-PD-1 antibody, anti-programmed death ligand 1 (PD-L1) antibody, CD19/CD3-bispecific antibody, and so on.
8. Confirmed evidence showing positiveness of anti-CD19 scFv reaction in patient serum.
9. Prior CD19 targeted therapy.
10. Prior CAR-T therapy or other genetically modified T cell therapy.
11. Presence of DSA directed against STAR T cells.
12. Patients who participated in other clinical trials within 4 weeks prior to enrollment.
13. Uncontrolled infectious diseases or other serious illnesses, including but not limited to infections [e.g., human immunodeficiency virus (HIV) infection or acute or chronic active hepatitis B (HBV) or C (HCV) infection], congestive heart failure, unstable angina, arrhythmias, or that pose an unpredictable risk in the opinion of the attending physician.
14. The presence of uncontrollable serous membrane fluid, such as massive pleural effusion or ascites.
15. A history of stroke or intracranial hemorrhage within 3 months prior to enrollment.
16. Major surgery or trauma occurred within 28 days prior to enrollment, or major side effects have not been recovered.
17. History of allergies to any of the ingredients in cell products.
18. Conditions in which a known mental or physical illness interferes with cooperation with the requirements of the study or disrupts the results or interpretation of the results and, in the opinion of the therapeutic investigator, makes the patient unfit for study participation.
19. There is the situation that the researcher's judgment will interfere with the whole study participation; Situations where there is significant risk to the subject; Or interferes with the interpretation of research data.
20. Inability to understand or unwillingness to sign informed consent.
21. Researchers believe that other reasons are not suitable for clinical trials.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-03-20 (Estimated); Primary Completion 2026-03-20 (Estimated); Study Completion 2027-03-20 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Incidence of Adverse Events (AEs) defined as DLT | 12 months
  DLT is defined as any AE related to the investigational drug that occurs within 28 days after administration of the STAR T cells and meets any one of the criteria listed in the DLT criteria. Cytokine release syndrome (CRS) and immune cell-associated neurotoxicity syndrome (ICANS) were graded according to American Society for Transplantation and Cellular Therapy (ASTCT) 2019 criteria. GvHD according to criteria defined by the Mount Sinai Acute GVHD International Consortium. Other AEs were graded according to common terminology criteria for adverse events (CTCAE) v5.0.
  * Grade 3 acute GVHD (aGVHD) that is not resolved to Grade 1 or 2 within 7 days, with the exception of isolated skin involvement aGVHD;
  * Grade 4 CRS or grade 3 CRS that is not resolved to grade 2 or lower within 2 weeks;
  * Grade 3 ICANS lasting for ≥7 days or Grade 4 ICANS;
  * Any other Grade ≥4 and Grade 3 AEs related to the STAR T that lasts for ≥14 days, except hematology toxicity.
Phase 1: RP2D | 12 months
  The RP2D was determined through phase 1 study.
Phase 2: Best objective Response Rate | 12 months
  The incidence of complete response (CR), partial response (PR), stable disease (SD), progressive disease (PD), or unevaluable (UE) as the best response to treatment assessed by investigators and based on the Lugano 2014 assessment criterion.

SECONDARY OUTCOMES:
Phase 2: Overall Survival (OS) | 12 months after the first infusion of CD19-STAR T cells
  OS is defined as the time from CD19-STAR T cells infusion to the date of death. Subjects who have not died by the analysis data cutoff date will be censored at their last contact date.
Phase 2: Progression Free Survival (PFS) | 12 months after the first infusion of CD19-STAR T cells
  PFS is defined as the time from the CD19-STAR T cells infusion date to the date of disease progression assessed by investigators and based on the Lugano 2014 assessment criterion, or death any cause. Participants not meeting the criteria for progression by the analysis data cutoff date were censored at their last evaluable disease assessment date.
Phase 2: Time to response (TTR) | 12 months
  TTR is defined as the time from CD19-STAR T infusion to first assessed CR or PR by investigators and based on the Lugano 2014 assessment criterion.
Phase 2: Duration of Response (DOR) | 12 months
  DOR is defined as the date of their first CR or PR (which is subsequently confirmed) to PD assessed by investigators and based on the Lugano 2014 assessment criterion for r/r B-cell NHL, or death regardless of cause.
Pharmacokinetics: Number and copy number of CD19-STAR T cells (phase 1 and phase 2) | 12 months
  Number and copy number of CD19-STAR T cells were assessed by number in peripheral blood. Blood samples were collected before and one year after cell infusion (until CD19-STAR T cells were not detected for two consecutive times) to detect the number and copy number of CD19-STAR T cells, and to evaluate the pharmacokinetics of CD19-STAR T.
Pharmacokinetics: Persistence of CD19-STAR T (phase 1 and phase 2) | 12 months
  Persistence of CD19-STAR T cell assessed by number in peripheral blood.
Pharmacodynamics: Peak level of cytokines in serum (phase 1 and phase 2) | Up to 28 days after infusion
  The cytokines mainly include interleukin-2 (IL-2 ), IL-6, IL-8, IL-10, tumor necrosis factor-α (TNF-α), C reactive protein (CRP), ferritin. Peak was defined as the maximum post-baseline level of the cytokine.

OTHER OUTCOMES:
Phase 1: Levels of donor-specific anti-HLA antibodies (DSA) in blood. | 12 months
  DSA refers to the specific antibody produced in the recipient's body targeting donor antigens after receiving STAR T cell infusion from healthy donors.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Biotherapeutic Department of Chinese PLA General Hospital, Beijing, Beijing Municipality
  - School of medicine, Tsinghua University & Changping Laboratory, Beijing

IPD SHARING:
Plan to Share IPD: No